CLINICAL TRIAL: NCT06011499
Title: Internet-Based Lifestyle Intervention to Eradicate Obese Frailty in Prostate Cancer Survivors (iLIVE)
Brief Title: Internet-Based Lifestyle Intervention to Eradicate Obese Frailty in Prostate Cancer Survivors, iLIVE
Acronym: iLIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Oregon Health and Science University (Other); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Kerri Winters, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00025281; R01CA275055 (NIH); NCI-2023-03141 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00025281 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors are blinded to participant group assignment after completing the baseline assessment and prior to randomization. Adverse events will be reviewed on a quarterly basis by the research team in a blinded fashion
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (iLIVE) (Experimental): Patients receive online access to an interactive weight loss website and participate in online group based resistance training sessions (iLIVE) on study. Patients also use a Fitbit fitness tracker and Aria smart scale while on study.
  Interventions: Other: Internet-Based Exercise Intervention; Other: Internet-Based Diet Intervention
- Arm II (usual care) (Active Comparator): Patients receive usual care with access to online survivorship and exercise recommendations and use a Fitbit fitness tracker and Aria (registered trademark) smart scale while on study.
  Interventions: Other: Education Intervention

INTERVENTIONS:
Other: Internet-Based Exercise Intervention — Participate in online supervised, group resistance training sessions (iLIVE)
  Arms: Arm I (iLIVE)
Other: Internet-Based Diet Intervention — Receive online access to an interactive website with a series of weekly self-directed and interactive sessions on various topics associated with diet and weight loss (iLIVE)
  Arms: Arm I (iLIVE)
Other: Education Intervention — Receive usual care receiving educational information about diet and exercise for cancer survivors
  Arms: Arm II (usual care)

SUMMARY:
This clinical trial tests the effectiveness of an online weight loss plus resistance training intervention (iLIVE) to decrease obesity and improve frailty in men with prostate cancer who received androgen deprivation therapy (ADT). Androgen deprivation therapy increases the risk of frailty, weight gain and obesity in prostate cancer survivors. The combination of frailty and obesity can lead to a decrease in quality of life and an increased risk of recurrent falls. Using iLIVE may improve obesity and frailty in men with prostate cancer who receive ADT.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To test the effectiveness of a combined online weight loss plus resistance training intervention (iLIVE) on obese frailty in prostate cancer survivors (PCS) on ADT.

SECONDARY OBJECTIVES:

I. To understand the effect of iLIVE on health behaviors, physical functioning, and quality of life II. To understand facilitators and barriers to implementing iLIVE in clinical and community practice

OUTLINE: Patients are randomized to arm I or II. Key stakeholders are identified for implementation outcomes

ARM I: Patients receive online access to an interactive weight loss website and participate in online group based resistance training sessions (iLIVE) on study. Patients also use a Fitbit fitness tracker and Aria (registered trademark) smart scale while on study.

ARM II: Patients receive usual care with access to online survivorship and exercise recommendations and use a Fitbit fitness tracker and Aria (registered trademark) smart scale while on study.

Patients are followed for 6 months after completion of intervention.

Key stakeholders complete an interview while on study to assess barriers and facilitators to implementation of iLIVE into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* INTERVENTION PARTICIPANTS: Age 18 or older
* INTERVENTION PARTICIPANTS: Diagnosed with histologically confirmed prostate cancer
* INTERVENTION PARTICIPANTS: Received >= 6 months of ADT any time in the past 10 years
* INTERVENTION PARTICIPANTS: Completed radiotherapy, chemotherapy and/or surgery > 6 weeks prior to
* INTERVENTION PARTICIPANTS: No intent to start adjuvant chemotherapy or radiotherapy within 6 months of enrollment
* INTERVENTION PARTICIPANTS: Overweight or obese (body mass index > 25 kg/m2 to BMI ≤ 50).
* INTERVENTION PARTICIPANTS: Evidence of frailty by meeting three or more of the following frailty criteria: weakness, slowness, fatigue, inactivity, and/or illness
* INTERVENTION PARTICIPANTS: Not currently engaging in structured diet or resistance strength training exercise program
* INTERVENTION PARTICIPANTS: Willing to be randomized into either study arm and adhere to study protocol
* INTERVENTION PARTICIPANTS: Home internet sufficient for videoconferencing
* INTERVENTION PARTICIPANTS: Signed informed consent
* IMPLEMENTATION PARTICIPANTS: Be a key stakeholder (i.e., healthcare provider or administrative, or intervention participant [completers, partial completers, or no participation])
* IMPLEMENTATION PARTICIPANTS: Verbal informed consent following receipt of an information sheet

Exclusion Criteria:

* INTERVENTION PARTICIPANTS: Unintentional weight loss > 5% within the last year
* INTERVENTION PARTICIPANTS: Contraindication to moderate intensity exercise
* INTERVENTION PARTICIPANTS: Health or medical condition that affects weight status/body composition (e.g., Cushing's syndrome, uncontrolled hyper-/hypo- thyroidism)
* INTERVENTION PARTICIPANTS: Active malignancy (other than non-melanoma skin cancer)
* INTERVENTION PARTICIPANTS: Not fluent in English and therefore incapable of answer survey questions, following directions during exercise or performance testing, and providing informed consent in English
* INTERVENTION PARTICIPANTS: Currently taking or have taken creatine supplement in the month preceding baseline creatine testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in overweight/obesity | At baseline, 3 months, 6 months and 12 months
  Measured from weight assessed on the Aria (registered trademark) scale at the time of the online assessment and self-reported height. Overweight is defined as body mass index > 25 kg/m^2 and a 5% loss will be viewed as a successful outcome.
Change in sarcopenia | At baseline and 6 months
  Measured by 30 mg D3 creatine (D3Cr) capsule which they will ingest and then urinate on a test strip on the second void upon waking 3-6 days later. The enrichment of D3Cr will be measured from the test strip along with urine creatine and creatinine. Will use a cutoff of < 10.75 kg/m^2 (moderate sarcopenia).
Change in slowness | At baseline, 3 months and 6 months
  Measured by the fastest time of two 4m walks at a usual pace administered by study staff by remote teleconference. Will use a cut point for "slowness" in older men of speed < 1.0 m/s - a clinically meaningful cutoff that predicts falls and loss of independence.
Change in weakness | At baseline, 3 months, and 6 months
  Measured by the seconds required to rise from a chair five times, administered by study staff by remote teleconference. Chair stand time > 12 seconds predicts a 2.4 increased risk of falls in older adults and we will apply this cutoff for "weakness."
Change in inactivity | At baseline, 3 months, 6 months, and 12 months
  Measured by physical activity-related energy expenditure, calculated from self-report on the 41-item Community Health Activities Model Program for Seniors (CHAMPS) physical activity questionnaire. We will use < 383 kcals per week spent in moderate-vigorous intensity activity as our low activity cut point. Measured also by Fitbit.
Change in frailty | At baseline, 3 months, 6 months, and 12 months
  Measured using the 4-item short form (SF)-36 Vitality Scale. Will use cut points of scores of < 50.00 (normed) for prostate cancer survivors (PCS) aged 50-64 years or scores less than 40.00 (normed) for PCS aged 65+ years.

SECONDARY OUTCOMES:
Change in health behaviors | At baseline, 3 months, 6 months, and 12 months
  Dietary intake measured using a 2-day diet recalls of 1-weekday and 1 weekend day will be collected by a registered dietitian via telephone and entered into the National Cancer Institute-developed Automated Self-Administered 24-hour. Physical activity measured using CHAMPS as described above. We will also assess free-living physical activity over 7-days using Fitbits.
Change in physical functioning | At baseline, 3 months, 6 months, 12 months
  Measured by Timed Up and Go using a widely used clinical measure of functional mobility that evaluates the time it takes to rise from a chair, walk 3m, turn around, and return and sit in the chair. SF-36 Physical Function measured using a 10-item physical function subscale of the SF-36.
Change in quality of life | At baseline, 3 months, 6 months, and 12 months
  Measured by European Quality of Life-5D with 1 question in 5 separate domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Scores will also be used to calculate Quality of Life Adjusted Years for cost-effectiveness analysis. Healthcare utilization measured using a brief questionnaire that assesses physician and emergency room visits, hospitalizations, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Winters-Stone, Principal Investigator — OHSU Knight Cancer Institute
Locations (2):
- United States (2):
  - University of Alabama, Birmingham, Alabama
  - OHSU Knight Cancer Institute, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
All individual quantitative participant data collected during the trial, after deidentification.
Time Frame: Beginning 3 months following final publication
Access Criteria: Access will be provided to investigators who provide a methodologically sound proposal and complete a data sharing agreement that includes commitments to: (1) using the data only for research purposes and not to identify any individual participant, (2) securing the data using appropriate computer technology, and (3) destroying or returning the data after analyses are completed.
  Proposals should be directed to wintersk@ohsu.edu. To gain access to data, data requestors will need to sign a data sharing agreement.